CLINICAL TRIAL: NCT00003762
Title: Randomized Phase II Study of Docetaxel and Gemcitabine for Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Docetaxel and Gemcitabine in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-982452; NCI-2012-02294 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000066887 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-05-02; First posted 2004-06-24 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I: docetaxel + gemcitabine (Experimental): Patients receive docetaxel IV over 1 hour on day 1 followed by gemcitabine IV over 30 minutes on days 1, 8, and 15. Patients continue treatment every 28 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with either stable disease or complete/partial response who discontinue treatment after 4-6 courses may be eligible for NCCTG-97-24-51.
  Quality of life is assessed before treatment and before each course of therapy.
  Patients are followed every 3 months for 1 year, then every 3 months for 5 years.
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride
- Arm II: docetaxel + gemcitabine (Experimental): Patients receive docetaxel IV over 1 hour and gemcitabine IV over 30 minutes on days 1 and 15. Patients continue treatment every 28 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with either stable disease or complete/partial response who discontinue treatment after 4-6 courses may be eligible for NCCTG-97-24-51.
  Quality of life is assessed before treatment and before each course of therapy.
  Patients are followed every 3 months for 1 year, then every 3 months for 5 years.
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride
- Arm III: docetaxel + gemcitabine (Experimental): Patients receive docetaxel IV on day 1 and gemcitabine IV on days 1, 8, and 15. Patients continue treatment every 28 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with either stable disease or complete/partial response who discontinue treatment after 4-6 courses may be eligible for NCCTG-97-24-51.
  Quality of life is assessed before treatment and before each course of therapy.
  Patients are followed every 3 months for 1 year, then every 3 months for 5 years.
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of two regimens of docetaxel plus gemcitabine in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate of patients with stage IIIB or IV nonsmall cell lung cancer to different schedules of docetaxel and gemcitabine therapy. II. Evaluate the toxicity of this treatment in these patients. III. Describe the quality of life parameters of patients receiving this combination therapy. IV. Determine the survival rate of these patients.

OUTLINE: This is a randomized study. Patients are stratified by disease (stage IIIB vs stage IV) and performance status (0 vs 1). Patients are randomized to one of two treatment arms (Arm I now closed). Arm I: Patients receive docetaxel IV over 1 hour on day 1 followed by gemcitabine IV over 30 minutes on days 1, 8, and 15. (closed as of 8/31/1999) Arm II: Patients receive docetaxel IV over 1 hour and gemcitabine IV over 30 minutes on days 1 and 15. Arm III: Patients receive docetaxel IV on day 1 and gemcitabine IV on days 1, 8, and 15. Patients continue treatment every 28 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients with either stable disease or complete/partial response who discontinue treatment after 4-6 courses may be eligible for NCCTG-97-24-51. Quality of life is assessed before treatment and before each course of therapy. Patients are followed every 3 months for 1 year, then every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 19-53 patients will be accrued for this study within 6-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IIIB/IV nonsmall cell lung cancer eligible for first line chemotherapy Measurable disease (must be outside radiation port or proof of progressive disease) Metastatic CNS disease allowed if treated and stable for at least 21 days prior to study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Greater than 12 weeks Hematopoietic: Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Absolute neutrophil count at least 1500/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) Alkaline phosphatase no greater than 3 times ULN AST no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: At least 3 months since prior myocardial infarction No uncontrolled congestive heart failure No uncontrolled arrhythmias Other: Not pregnant or nursing Fertile patients must use effective contraception Peripheral neuropathy less than grade 2 No history of hypersensitivity to products containing polysorbate 80 No other significant medical condition No meningeal carcinomatosis No weight loss of greater than 10% within past 3 months due to disease

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy to pelvis, spine, or long bones and recovered No prior radiotherapy to at least 30% of bone marrow Surgery: Greater than 4 weeks since prior major surgery Other: At least 3 weeks since prior investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 1999-02; Primary Completion 2003-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota

REFERENCES:
- [Background] Huschka MM, Mandrekar SJ, Schaefer PL, Jett JR, Sloan JA. A pooled analysis of quality of life measures and adverse events data in north central cancer treatment group lung cancer clinical trials. Cancer. 2007 Feb 15;109(4):787-95. doi: 10.1002/cncr.22444. PMID 17211864
- [Background] Jatoi A, Hillman S, Stella P, Green E, Adjei A, Nair S, Perez E, Amin B, Schild SE, Castillo R, Jett JR; North Central Cancer Treatment Group. Should elderly non-small-cell lung cancer patients be offered elderly-specific trials? Results of a pooled analysis from the North Central Cancer Treatment Group. J Clin Oncol. 2005 Dec 20;23(36):9113-9. doi: 10.1200/JCO.2005.03.7465. PMID 16361618